CLINICAL TRIAL: NCT00115063
Title: Loss - Louisiana Obese Subjects Study
Brief Title: LOSS- Louisiana Obese Subjects Study
Acronym: LOSS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: ethical issues of continuing control group without treatment
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Louisiana Office of Group Benefits (Unknown)
Responsible Party: Principal Investigator, Donna H. Ryan, MD, Professor, Adjunct, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 25002
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Results first posted 2010-06-07 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: obesity; Low Calorie Diet; Obesity Pharmacotherapy; Pragmatic Clinical Trial
MeSH Terms: conditions — Obesity | interventions — sibutramine; Orlistat; Diethylpropion; Caloric Restriction; One Health; Adiposity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intensive Medical Intervention including Low Calorie Liquid Diet, Weight loss medications, Group Behavioral Therapy and a "Tool Box" approach
  Interventions: Behavioral: group sessions; Drug: sibutramine, orlistat, diethylpropion; Behavioral: Low Calorie Diet, Health One; Other: Intensive Medical Combination Therapy for Obesity
- 2 (Active Comparator): Access to Weight Loss Informational Website sponsored by the Mayo Clinic
  Interventions: Other: Control Condition

INTERVENTIONS:
Behavioral: group sessions — group sessions lead by a trained primary care clinic employee
  Arms: 1
Drug: sibutramine, orlistat, diethylpropion — dosage modified according to package insert instructions at discretion of primary care physicians
  Arms: 1
Behavioral: Low Calorie Diet, Health One — liquid diet for 8-12 weeks to induce weight loss
  Arms: 1
Other: Intensive Medical Combination Therapy for Obesity — Very Low Calorie Liquid diet, Group Behavioral Therapy, Meal Replacement Therapy, Obesity Pharmacotherapy and a "Treatment Toolbox".
  Arms: 1
Other: Control Condition — Access to the Mayo Clinic weight management website and usual care from the primary care physician
  Arms: 2

SUMMARY:
LOSS is a pragmatic clinical evaluation of intensive medical approaches to weight loss for individuals with extreme obesity (body mass index [BMI] 40-60 kg/m2). The intensive medical treatment is designed to produce 25% weight loss from baseline and to maintain at least 20% weight loss from baseline. The intensive medical treatment is compared to a usual care treatment model where individuals utilize self directed approaches to weight loss. The active treatment period is three years, followed by two years of observation.

DETAILED DESCRIPTION:
LOSS is a pragmatic clinical trial designed to evaluate intensive medical treatment for patients with severe obesity who would otherwise qualify as candidates for obesity surgery and who are covered by the Louisiana Office of Group Benefits (OGB) Health Insurance. LOSS will track the efficacy, safety and costs to compare two patient management approaches - intensive medical treatment, or a usual medical care treatment model. Recruitment will be done by mailers to insured patients to identify eligible candidates. We will randomly assign eligible volunteers to intensive medical treatment (n=240) or usual care (n=240). Patients will be evaluated annually and medical treatments are given in eight clinics around Louisiana. The eight sites are in Alexandria, Baton Rouge, Lafayette, Lake Charles, Monroe, Hammond, New Orleans and Shreveport.

Hypothesis:

We hypothesize that we can achieve weight loss after two and five years that exceeds 20% from baseline with intensive medical management of persons with class III obesity and that this weight loss is greater than that achieved with usual medical care including access to a weight management web site.

Our secondary hypotheses are: 1) that the weight loss at year 2 and 5 in the intensive medical group is associated with improvements in blood pressure, fasting glucose, lipids, health-related quality of life and psychosocial measures and is greater improvement than that achieved with usual medical care and access to a website; and 2) that total medical costs in the intensive medical management group will compare favorably to total medical costs in the usual care group (i.e., total reimbursement from insurance costs will be less, even when the expense of the treatment is considered).

Overall Aim:

The overarching aim of this study is to observe the effect of an intensive medical management program versus usual care for class III obesity on weight loss, total medical costs and, on measures of health risks associated with weight loss (blood pressure, blood glucose, blood lipids, and health-related quality of life).

Specific Aims:

Primary: The primary specific aim of the LOSS study is to test the hypothesis that the weight loss efficacy at years 2 and 5 for an intensive medical treatment program for Class III obesity produces greater weight loss, as compared to a condition of usual care.

Secondary: The secondary aims of the study are:

* To evaluate the percent change in body weight, absolute change in body weight (kilograms) and percent excess weight lost from baseline at months 3, 6, 12, 24, 36, 48 and 60 for medically treated patient groups, and at years 1, 2, 3, 4 and 5 for both groups.
* To evaluate the number and proportion of subjects who maintain 100% and 80% of 12 months weight lost at months 24, 36, 48 and 60 for medically treated patients and at years 2, 3, 4 and 5 for both groups.
* To evaluate the changes from baseline in blood pressure, pulse rate, and efficacy laboratory parameters at visits on months 3, 6, 12, 24, 36, 48 and 60 for the medically treated patient group, and at years 1, 2, 3, 4 and 5 for both groups.
* To assess the safety and tolerability of the intervention regimens at months 3, 6, 12, 24, 36, 48 and 60 for the medically treated patient group.
* To assess the total medical costs of the participants treated with intensive medical treatment and for the patients receiving usual care at years 1, 2, 3, 4 and 5.
* To assess additional psychosocial and economic measures (health-related quality of life, pain, depression, and stress) for the intervention group at months 4, 8, 12, 24, 36, 48 and 60 months for both groups at years 1, 2, 3, 4, and 5.
* To compare subgroups of patients with class III obesity to determine if differences in outcome exist for gender, race, education level, decades of age and presence of co-morbid conditions.

The Pennington Biomedical Research Center is the lead institution for the project. Pennington Management of Clinical Trials (PMCT) will serve as the Coordinating Center to manage enrollment and data acquisition and will report all data of health and cost results to a Data Safety Monitoring Board on a regular basis. Major data reports and scientific publications occur at years 2 and 5.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the Exclusive Provider Organization (EPO), Managed Care Organization (MCO) and Preferred Provider Organization (PPO) programs of the Louisiana State Employees Group Benefits Health Insurance
* Agree to travel for treatment to the assigned study site
* Agree to randomized treatment assignment
* Male and females age 20-60 years
* Body Mass Index >40kg/m2 but < 60 kg/m2
* Females must be non-pregnant and using an approved contraception method
* Complete Blood Count (CBC): normal hematocrit, white count and platelet count, unless waived by Principal Investigator (PI)
* Uric Acid <9.0 mg/dl
* Normal Creatinine
* Normal Thyroid Stimulating Hormone (TSH)
* Negative urine pregnancy test for women of childbearing potential
* Able to give written informed consent
* Able to comply with study procedures

Exclusion Criteria:

Factors that may limit adherence to interventions or affect conduct of the trial:

* Unable or unwilling to give informed consent or communicate with local study staff
* Hospitalization for psychiatric illness or substance use/abuse within the past year
* Self-report of alcohol or substance abuse within the past twelve months
* Current major depressive episode or history of suicidal behaviors
* Endorsement of significant recent suicidal ideation (as determined by PI)
* Travel plans that do not permit participation
* History of prior bariatric surgery, small bowel resection, or extensive bowel resection
* Current use of chronic systemic corticosteroids, appetite suppressants, antipsychotic medication, herbal medications for weight loss or any medication not approved by the PI.
* Another member of the household is a participant or staff member in the study
* History of eating disorder such as anorexia nervosa, bulimia, or binge eating
* Diagnosis of schizophrenia, other psychotic disorders, bipolar disorder, or personality disorder (as determined by the PI)
* Currently pregnant or nursing or plans to become pregnant in the next five years
* Except for non-melanoma skin cancer, cancer requiring treatment in the past five years, unless the prognosis is excellent
* Self report of Human Immunodeficiency Virus (HIV) positive, hepatitis C or active tuberculosis
* Cardiovascular disease event within the past year
* Severe congestive heart failure (New York Heart Association [NYHA] Functional Class III, IV)
* Second degree or greater heart block
* Blood Pressure >160 systolic or >100 diastolic on two consecutive visits, unless treated and re-screened
* Based upon responses to psychological screening or an interview, patients may be excluded by the study psychologist.
* Other medical, psychiatric, or behavioral limitations that in the judgment of the investigator may interfere with study participation or the ability to follow the intervention protocol.
* Pregnancy is to be avoided during the study. Women who have not had a hysterectomy or oophorectomy must have a negative urine pregnancy test result at screening. Women of childbearing potential will be allowed to participate if they have undergone tubal ligation, or use one of the following types of contraception: properly used condom or diaphragm, oral contraceptives, hormonal implant, or intrauterine device (IUD). Sexual abstinence may constitute an acceptable birth control method for this study with investigator approval. Women with male partners who have had a successful vasectomy (more than one year of unprotected sexual intercourse without pregnancy) are not required to use additional birth control methods as long as the relationship remains exclusive, and the woman agrees to use an approved contraception method with any other male partner. Questions regarding individual patient contraceptive practices should be directed to the Principal Investigator.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 390 (Actual)
Dates: Start 2005-07; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna H Ryan, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Management of Clinical Trials, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Johnson WD, Brashear MM, Gupta AK, Rood JC, Ryan DH. Incremental weight loss improves cardiometabolic risk in extremely obese adults. Am J Med. 2011 Oct;124(10):931-8. doi: 10.1016/j.amjmed.2011.04.033. PMID 21962313
- [Derived] Ryan DH, Johnson WD, Myers VH, Prather TL, McGlone MM, Rood J, Brantley PJ, Bray GA, Gupta AK, Broussard AP, Barootes BG, Elkins BL, Gaudin DE, Savory RL, Brock RD, Datz G, Pothakamuri SR, McKnight GT, Stenlof K, Sjostrom LV. Nonsurgical weight loss for extreme obesity in primary care settings: results of the Louisiana Obese Subjects Study. Arch Intern Med. 2010 Jan 25;170(2):146-54. doi: 10.1001/archinternmed.2009.508. PMID 20101009
- See also: Pennington Biomedical Research Center home page — http://www.pbrc.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive Medical Intervention: Intensive Medical Intervention including Low Calorie Liquid Diet, Weight loss medications, Group Behavioral Therapy and a "Tool Box" approach
- Access to Weight Loss Informational Website: Access to Weight Loss Informational Website sponsored by the Mayo Clinic
Period: Overall Study
Arm/Group | Intensive Medical Intervention | Access to Weight Loss Informational Website
Started | 200 | 190
Completed | 101 | 86
Not Completed | 99 | 104
Not completed — Lost to Follow-up | 98 | 104
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Medical Intervention | Access to Weight Loss Informational Website | Total
Number analyzed (Participants) | 200 | 190 | 390
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 200 | 190 | 390
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (0.6) | 47.1 (0.6) | 47.2 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 159 | 326
  Male | 33 | 31 | 64
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 0 | 1
  White | 149 | 147 | 296
  Black or African American | 50 | 43 | 93
Region of Enrollment [Number; unit: participants]
  United States | 200 | 190 | 390

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline Weight
Time Frame: Baseline, 2 years
Population: This analysis was done on the completers, those that completed the 2 year study visit.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Intensive Medical Intervention | Access to Weight Loss Informational Website
Number analyzed (Participants) | 101 | 86
Percent change | -9.7 (1.3) | -0.4 (0.7)
Statistical Analysis 1: Comparison: Intensive Medical Intervention vs Access to Weight Loss Informational Website; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Change in Weight From Baseline in Kilograms (kg)
Time Frame: Baseline, 2 years
Population: This analysis was done on the completers, those that completed the 2 year study visit.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Intensive Medical Intervention | Access to Weight Loss Informational Website
Number analyzed (Participants) | 101 | 86
kg | -12.7 (1.7) | -0.5 (0.9)
Statistical Analysis 1: Comparison: Intensive Medical Intervention vs Access to Weight Loss Informational Website; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Change in Blood Pressure
Time Frame: Baseline, 2 years
Population: This analysis was done on the completers, those that completed the 2 year study visit.
Measure: Mean (Standard Error); unit: millimeter of mercury (mm Hg)
Arm/Group | Intensive Medical Intervention | Access to Weight Loss Informational Website
Number analyzed (Participants) | 101 | 86
millimeter of mercury (mm Hg)
  systolic blood pressure | -14.7 (2.4) | -8.6 (2.6)
  dystolic blood pressure | -4.4 (1.8) | -3.2 (1.5)
Statistical Analysis 1: Comparison: Intensive Medical Intervention vs Access to Weight Loss Informational Website; Test type: Superiority or Other; p = 0.09, t-test, 2 sided — P-value for systolic blood pressure mean
Statistical Analysis 2: Comparison: Intensive Medical Intervention vs Access to Weight Loss Informational Website; Test type: Superiority or Other; p = 0.60, t-test, 2 sided — P-value for dystolic blood pressure mean

4. Secondary Outcome: Percent Change in Blood Tests- Low Density Lipoprotein (LDL), High Density Lipoprotein (HDL), Triglycerides and Uric Acid
Time Frame: Baseline, 2 years
Population: This analysis was done on the completers, those that completed the 2 year study visit.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Intensive Medical Intervention | Access to Weight Loss Informational Website
Number analyzed (Participants) | 101 | 86
Percent change
  LDL | 1.8 (2.4) | 0.7 (2.4)
  HDL | 7.9 (1.8) | 1.5 (1.8)
  Triglycerides | -9.2 (3.5) | -4.8 (4.3)
  Uric Acid | -3.0 (2.4) | 3.1 (1.8)
Statistical Analysis 1: Comparison: Intensive Medical Intervention vs Access to Weight Loss Informational Website; Test type: Superiority or Other; p = 0.73, t-test, 2 sided — P-value for LDL cholesterol
Statistical Analysis 2: Comparison: Intensive Medical Intervention vs Access to Weight Loss Informational Website; Test type: Superiority or Other; p = 0.01, t-test, 2 sided — P-value for HDL cholesterol
Statistical Analysis 3: Comparison: Intensive Medical Intervention vs Access to Weight Loss Informational Website; Test type: Superiority or Other; p = 0.42, t-test, 2 sided — P-value for triglycerides
Statistical Analysis 4: Comparison: Intensive Medical Intervention vs Access to Weight Loss Informational Website; Test type: Superiority or Other; p = 0.05, t-test, 2 sided — P-value for uric acid

5. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) in Milligrams Per Deciliter (mg/dL)
Time Frame: Baseline, 2 years
Population: This analysis was done on the completers, those that completed the 2 year study visit.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Intensive Medical Intervention | Access to Weight Loss Informational Website
Number analyzed (Participants) | 101 | 86
mg/dL | 2.4 (2.1) | 6.7 (2.1)
Statistical Analysis 1: Comparison: Intensive Medical Intervention vs Access to Weight Loss Informational Website; Test type: Superiority or Other; p = 0.16, t-test, 2 sided

6. Secondary Outcome: Change in Duke Activity Status Index (DASI) Questionnaire Score
Description: The DASI was used to access changes in fuctional capacity during the study. The highest score possible is 58.2 and the lowest is 0. The score for each individual question varied depending on the intensity of the activity being evaluated. The higher the score, the more physically active a person is to this set of activities of daily living questions.
Time Frame: Baseline, 2 years
Population: This analysis was done on the completers, those that completed the 2 year study visit.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intensive Medical Intervention | Access to Weight Loss Informational Website
Number analyzed (Participants) | 101 | 86
units on a scale | -2.1 (1.7) | -11.6 (2.0)
Statistical Analysis 1: Comparison: Intensive Medical Intervention vs Access to Weight Loss Informational Website; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected at all study visits for both groups from study start to 2 years.
Description: Only serious adverse events were tracked for this study.
Arm/Group | Intensive Medical Intervention | Access to Weight Loss Informational Website
Serious Adverse Events (participants affected / at risk) | 20/200 | 8/190
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Medical Intervention (N=200) | Access to Weight Loss Informational Website (N=190)
Hernia repair (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hospitalization for coronary stent replacement (Vascular disorders) | 1 (1) | 0 (0)
Hospitalization for deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Surgery for cyctocele (Renal and urinary disorders) | 1 (1) | 0 (0)
Surgical incision and drainage of abscess (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalization for pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization for hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) — Patient had history of mental illness
Hospitalization for arm fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hospitalization for nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hospitalization for asthma and bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest heaviness (Cardiac disorders) | 1 (1) | 0 (0) — Referred to cardiologist
Elevated blood pressure and mood swings (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 2 (2) | 0 (0) — One patient reported chest pain and underwent a angiograpy, results were normal. A second patient reported chest pain and was hospitalized, diagnosed with dehydration.
Cervical disk surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bleeding duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (Cardiac disorders) | 1 (1) | 0 (0) — Due to myocardial infarction
Total knee replacement surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
New-onset atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization for acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pacemaker insertion procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Hospitalization for back surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hospitalization for hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hospitalization for stent placement (Surgical and medical procedures) | 0 (0) | 1 (1)
Hysterectomy (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was stopped prematurely for efforts to be focused on assisting the Office of Group Benefits (OGB) in translating a policy that would allow for physician certification in order to offer participants the intensive treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No